CLINICAL TRIAL: NCT03560349
Title: A Multicenter Double Blinded Randomized Controlled Trial of the Efficacy of the Sphenopalatine Ganglion Block for the Treatment of the Postdural Puncture Headache After Labor Epidural
Brief Title: RCT of SPG Blocks for Post-dural Headache
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Both Study PI's left the institution
Sponsor: University of Utah (Other)
Collaborators: University of Colorado, Denver (Other); University of California, San Francisco (Other); Duke University (Other); Mayo Clinic (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110257
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Experimental): Transnasal blockade of SPG approach involving the application of 2 cc (approximately the size of a pea) of 2% lidocaine jelly on a cotton swab directed posteriorly towards the SPG in the nasal passage bilaterally. Cotton swab will be inserted to the back of the nasal passage until it can no longer be inserted any further. The cotton swab should remain in place for 15 minutes on both sides simultaneously. The patient will be instructed on how to perform this procedure on themselves, and they will be given supplies for a 7-day supply of medication to be administered two times per day at approximately 12 hour intervals.
  Interventions: Drug: Lidocaine HCl Gel 2%
- Placebo (Placebo Comparator): Transnasal blockade of SPG approach involving the application of 2 cc (approximately the size of a pea) of nasal saline jelly on a cotton swab directed posteriorly towards the SPG in the nasal passage bilaterally. Cotton swab will be inserted to the back of the nasal passage until it can no longer be inserted any further. The cotton swab should remain in place for 15 minutes. The patient will be instructed on how to perform this procedure on themselves, and they will be given supplies for a 7-day supply of medication to be administered up to two times per day at approximately 12 hour intervals.
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: Lidocaine HCl Gel 2% — Patients will be prescribed a regimen of 1 g acetaminophen q 8hrs alternating with 600 mg ibuprofen q 6 hours. In addition they will be instructed to continue oral fluid hydration and minimal activity for 24 hours.
  At 2-hours following the SPG blockade an EBP will be offered to patients. Patient will also be informed that they can request an EBP at any time. The SPG blockade will be performed twice daily in the hospital and twice daily at home, by the patient. The patient will also be informed, if that at anytime, they would like an EBP, it can be provided.
  While the study is being conducted, patients will not be offered a SPG block unless enrolled in the study.
  Arms: Lidocaine
Drug: placebo gel — Patients will be prescribed a regimen of 1 g acetaminophen q 8hrs alternating with 600 mg ibuprofen q 6 hours. In addition they will be instructed to continue oral fluid hydration and minimal activity for 24 hours.
  At 2-hours following the SPG blockade an EBP will be offered to patients. Patient will also be informed that they can request an EBP at any time. The SPG blockade will be performed twice daily in the hospital and twice daily at home, by the patient. The patient will also be informed, if that at anytime, they would like an EBP, it can be provided.
  While the study is being conducted, patients will not be offered a SPG block unless enrolled in the study.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the effectiveness of the SPG block with lidocaine vs. SPG block with placebo on preventing the need for EBP in women who develop PDPH after accidental dural puncture during placement of LEA for labor.

DETAILED DESCRIPTION:
The postdural puncture headache (PDPH) is a well-documented complication of dural puncture. Depending on a number of factors, the overall incidence of PDPH following unintended dural puncture with an epidural placement needle is typically around 50%, but can be as high as 70% for certain populations.(1, 2, 3)

The headache is characterized by being frontal or occipital in nature, with a typical onset of 6-72 hours after dural puncture. It is normally exacerbated by the upright position and improved by the supine position. Associated symptoms may include photophobia, nausea, vomiting, dizziness, tinnitus, neck stiffness, decreased hearing and visual changes. (2) These symptoms tend to be extremely debilitating in affected patients, severely limiting their functional capacity until the resolution of the headache.(2) The compromise is even greater when considering these women also need to care for a newborn, as the time after birth is important for forming attachment and encompasses many new obligations for the new mother.

The treatment of the PDPH often begins with conservative treatment including supportive therapies such as hydration, bed rest, acetaminophen, NSAIDs, and oral opioids. In addition, some evidence exists for the use of caffeine (1,2). While these do not hasten recovery, they may improve symptoms. For PDPH of all etiologies, 72% will resolve spontaneously in 7 days and 89% by 14 days. (1)

For patients with moderate to severe symptoms or long lasting headaches, the gold standard for treatment of headaches that do not resolve is the epidural blood patch (EBP) (1,2,4). This treatment has been shown to be effective in 70-98% of patients (1,2,4). However, it has numerous contraindications including: fever, infection, coagulopathy, active neurological disease, patient refusal. In addition, a potential complication is yet another dural puncture. Also, while the EBP is generally very safe, it is an invasive procedure with its own complications; it has been associated with very rare but serious complications including: moderate long-lasting backache, meningitis, epidural abscess formation, epidural hematoma formation, and neurologic deficit development. (5-8)

The sphenopalatine ganglion (SPG) is a parasympathetic ganglion with fibers that innervate the cerebral and meningeal blood vessels cause vasodilation and activation of nociceptive fibers in the meninges, which is perceived as referred pain from the head by the sensory cortex. (9) So blockade of these fibers can theoretically relieve headache symptoms from other causes. The SPG block has been safely used for many years to treat chronic facial or head pain from cluster headaches, trigeminal neuralgia, postherpetic neuralgia, atypical facial pain from cancer, and CRPS I and II. (9)

The SPG block is safe and easy to perform. The only contraindications include patient refusal, a true allergy to local anesthetic, and Hereditary Hemorrhagic Telangiectasia (HHT). (9,10) Documented potential complications include transient nausea and epistasis. (9,10) The SPG is located in the pterygopalatine fossa, which is just posterior to the middle turbinate, and anterior to the pterygoid canal. It is about 5 mm in size and there is a 1 to 1.5 mm-thick layer of connective tissue and mucous membrane surrounding the ganglion, so drug enters easily by a topical application. (9-11) There are multiple approaches to the blockade of this ganglion, but the easiest and least invasive is the transnasal approach involving entering the nare with the application of lidocaine jelly on a cotton swab directed posteriorly in the nasal passage to the SPG. (9) The cotton swab should remain in place for 10 minutes. (9,10)

Recently, the SPG block has also been shown to be effective in relieving the symptoms of the PDPH in case series and case reports. One case series performed SPG blocks in 3 parturients with confirmed PDPH in the emergency room using 2% viscous lidocaine. All 3 patients had good relief after the intervention and did not require EPB. The authors suggested that the procedure can be safely and accurately performed in the emergency room, which will reduce visit time, provide good pain relief, and the EBP can be deferred. (10) Another case series of 32 patients with confirmed PDPH of multiple etiologies showed that the SPG block prevented the need for EBP in 69% of the cases. (12)

In addition, a recent randomized placebo controlled trial of SPG block vs. saline for acute headache in the ER showed that for patients with acute anterior headache, SPG block with bupivacaine resulted in a reduction of HA symptoms. However, reduction of headache symptoms was also seen in the SPG block with saline group, indicating a possible placebo effect of the performance of the block. (13)

The purpose of the study is to assess the effectiveness of the SPG block with lidocaine vs. SPG block with placebo on preventing the need for EBP in women who develop PDPH after accidental dural puncture during placement of LEA for labor.

ELIGIBILITY:
Inclusion Criteria:

* Females
* age 18-50
* Post Dural Puncture Headache after documented accidental dural puncture during placement of LEA for labor and no better explanation for headache
* onset of HA within 72 hours of delivery.

Exclusion Criteria:

* true allergy to local anesthesia
* Hereditary Hemorrhagic Telangiectasia
* inability to understand pain scores and other questionnaires
* inability to speak English
* contraindication to acetaminophen or NSAIDs
* temperature >38.5 C
* prior Epidural Blood Patch done for this headache

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Studying post partum women
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Epidural Blood Patch | 7 days after treatment with lidocaine or placebo block
  Proportion of postpartum women with a postdural puncture headache (PDPH) requesting epidural blood patch (EBP)

SECONDARY OUTCOMES:
Verbal Numerical Pain | 30 minutes, 1 hour, 2, hour, 1 day, 2, days, 3 days, 4 days, 5 days, 6 days, and 7 days after treatment with lidocaine or placebo block
  Verbal Numerical Pain score (0-10)
Verbal Functionality Score | 1 day, 2, days, 3 days, 4 days, 5 days, 6 days, and 7 days after treatment with lidocaine or placebo block
  Daily Questionnaire regarding functionality

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Background] Amorim JA, Gomes de Barros MV, Valenca MM. Post-dural (post-lumbar) puncture headache: risk factors and clinical features. Cephalalgia. 2012 Sep;32(12):916-23. doi: 10.1177/0333102412453951. Epub 2012 Jul 27. PMID 22843225
- [Background] Flaatten H, Rodt S, Rosland J, Vamnes J. Postoperative headache in young patients after spinal anaesthesia. Anaesthesia. 1987 Feb;42(2):202-5. doi: 10.1111/j.1365-2044.1987.tb03001.x. PMID 3826597
- [Background] Abouleish E, Vega S, Blendinger I, Tio TO. Long-term follow-up of epidural blood patch. Anesth Analg. 1975 Jul-Aug;54(4):459-63. doi: 10.1213/00000539-197554040-00012. PMID 125053
- [Background] Cornwall RD, Dolan WM. Radicular back pain following lumbar epidural blood patch. Anesthesiology. 1975 Dec;43(6):692-3. doi: 10.1097/00000542-197512000-00023. No abstract available. PMID 127535
- [Background] Mehta SP, Keogh BP, Lam AM. An epidural blood patch causing acute neurologic dysfunction necessitating a decompressive laminectomy. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):78-80. doi: 10.1097/AAP.0000000000000025. PMID 24310044
- [Background] Reynolds AF Jr, Hameroff SR, Blitt CD, Roberts WL. Spinal subdural epiarachnoid hematoma: a complication of a novel epidural blood patch technique. Anesth Analg. 1980 Sep;59(9):702-3. No abstract available. PMID 7191232
- [Background] Sperry RJ, Gartrell A, Johnson JO. Epidural blood patch can cause acute neurologic deterioration. Anesthesiology. 1995 Jan;82(1):303-5. doi: 10.1097/00000542-199501000-00038. No abstract available. PMID 7832316
- [Background] Nair AS, Rayani BK. Sphenopalatine ganglion block for relieving postdural puncture headache: technique and mechanism of action of block with a narrative review of efficacy. Korean J Pain. 2017 Apr;30(2):93-97. doi: 10.3344/kjp.2017.30.2.93. Epub 2017 Mar 31. PMID 28416992
- [Background] Kent S, Mehaffey G. Transnasal sphenopalatine ganglion block for the treatment of postdural puncture headache in obstetric patients. J Clin Anesth. 2016 Nov;34:194-6. doi: 10.1016/j.jclinane.2016.04.009. Epub 2016 May 11. PMID 27687372
- [Background] Kent S, Mehaffey G. Transnasal sphenopalatine ganglion block for the treatment of postdural puncture headache in the ED. Am J Emerg Med. 2015 Nov;33(11):1714.e1-2. doi: 10.1016/j.ajem.2015.03.024. Epub 2015 Mar 14. No abstract available. PMID 25819208
- [Background] Cohen S, Ramos D, Grubb W, Mellender S, Mohiuddin A, Chiricolo A. Sphenopalatine ganglion block: a safer alternative to epidural blood patch for postdural puncture headache. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):563. doi: 10.1097/AAP.0000000000000172. No abstract available. PMID 25340493
- [Background] Schaffer JT, Hunter BR, Ball KM, Weaver CS. Noninvasive sphenopalatine ganglion block for acute headache in the emergency department: a randomized placebo-controlled trial. Ann Emerg Med. 2015 May;65(5):503-10. doi: 10.1016/j.annemergmed.2014.12.012. Epub 2015 Jan 7. PMID 25577713